CLINICAL TRIAL: NCT00874549
Title: A Safety and Immunogenicity Evaluation of a Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) and a Meningococcal Polysaccharide Vaccine Groups A, C, Y, and W-135 Combined (Menomune® - A/C/Y/W-135) in Subjects 56 Years of Age or Older
Brief Title: Exploratory Trial to Evaluate the Safety and Immunogenicity of Menactra® and Menomune® Vaccines in Subjects ≥ 56 Years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA29
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Results first posted 2010-03-25 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Meningococcal Infections; Meningococcal Meningitis
Keywords: Meningococcal Vaccine; Menactra®; Menomune®
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Menomune Day 0 (Active Comparator): Participants received a single dose of Menomune® vaccine on Day 0.
  Interventions: Biological: Menomune®: A, C, Y, W-135 Meningococcal Polysaccharide
- Group 2: Menactra® Day 0 x 2 (Experimental): Participants received two single-dose injections of Menactra® vaccine on Day 0
  Interventions: Biological: Menactra®: Polysaccharide Diphtheria Toxoid Conjugate
- Group 3: Menactra® Day 0 and 14 (Experimental): Participants received a single dose of Menactra® vaccine on Day 0 and on Day 14
  Interventions: Biological: Menactra®: Polysaccharide Diphtheria Toxoid Conjugate
- Group 4: Menactra® Day 0 and 28 (Experimental): Participants received a single dose of Menactra® vaccine on Day 0 and on Day 28.
  Interventions: Biological: Menactra®: Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Menomune®: A, C, Y, W-135 Meningococcal Polysaccharide — 0.5 mL, Subcutaneous
  Other Names: Menomune®
  Arms: Group 1: Menomune Day 0
Biological: Menactra®: Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Group 2: Menactra® Day 0 x 2
Biological: Menactra®: Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL. Intramuscular
  Other Names: Menactra®
  Arms: Group 3: Menactra® Day 0 and 14
Biological: Menactra®: Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Group 4: Menactra® Day 0 and 28

SUMMARY:
Safety:

To describe the rates of immediate reactions, solicited injection-site and systemic reactions, all unsolicited adverse events, and serious adverse events following vaccination with either Menactra® vaccine or Menomune® vaccine.

Immunogenicity:

To evaluate the immune response to serogroups A, C, Y, and W-135 in each of the four study groups.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory and healthy, as determined by medical history.
* 56 years of age or older at the time of vaccination.
* Signed Institutional Review Board (IRB)-approved informed consent form.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman, inability to become pregnant or a negative urine pregnancy test at the time of enrollment.

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Serious chronic disease (i.e., cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric, etc) that is unstable or that might 1) interfere with the ability to participate fully in the study or 2) interfere with evaluation of the vaccines.
* Known or suspected impairment of immunologic function.
* Febrile illness within the last 72 hours or an oral temperature ≥ 100.4ºF at the time of inclusion.
* History of documented invasive meningococcal disease or previous meningococcal vaccination.
* Known or suspected receipt of a diphtheria-containing vaccine within the preceding 2 years.
* Administration of immune globulin or other blood products within the last three months, or injected or oral corticosteroids or other immunomodulator therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Systemic antibiotic therapy within the 72 hours prior to collection of any blood samples.
* Received any vaccine in the 28-day period prior to enrollment or scheduled to receive any vaccination through Visit 2 for Groups 1 and 2 and through Visit 3 for Groups 3 and 4. Influenza vaccines may be received 2 weeks before or after a study vaccination.
* Suspected or known hypersensitivity to latex or to any of the components of either Menactra® vaccine or Menomune® vaccine.
* Previous personal history of Guillain-Barré syndrome.
* Not available for the entire study period or unable to attend the scheduled visits or to comply with the study procedures.
* In females of childbearing potential, a positive or equivocal urine pregnancy test at enrollment.
* A nursing mother.
* Participation in another interventional clinical trial in the 4 weeks preceding enrollment or planning to participate in another interventional clinical trial during the planned period of this study.
* Current use of alcohol or recreational drugs that may interfere with the subject's ability to comply with trial visits or procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (6):
- United States (6):
  - Scottsdale, Arizona
  - Bardstown, Kentucky
  - Albuquerque, New Mexico
  - West Jordon, Utah
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 10 October 2007 to 25 August 2008 at 6 US clinical centers.
Pre-assignment Details: A total of 216 participants who met the inclusion and exclusion criteria were enrolled, vaccinated, and included in the analyses.
Groups:
- Group 1: Menomune® Day 0: Participants with no prior meningococcal vaccine exposure who had received no diphtheria-containing vaccine in the prior 2 years received a single dose of Menomune® subcutaneously on Day 0.
- Group 2: Menactra® Day 0 x 2: Participants with no prior meningococcal vaccine exposure who had received no diphtheria-containing vaccine in the prior 2 years received 2 single-dose injections of Menactra® intramuscularly on Day 0.
- Group 3: Menactra® Day 0 and 14: Participants with no prior meningococcal vaccine exposure who had received no diphtheria-containing vaccine in the prior 2 years received a single dose of Menactra® intramuscularly on Day 0 and again on Day 14.
- Group 4: Menactra® Day 0 and 28: Participants with no prior meningococcal vaccine exposure who had received no diphtheria-containing vaccine in the prior 2 years received a single dose of Menactra® intramuscularly on Day 0 and again on Day 28.
Period: Overall Study
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Started | 51 | 56 | 51 | 58
Completed | 50 | 55 | 47 | 56
Not Completed | 1 | 1 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28 | Total
Number analyzed (Participants) | 51 | 56 | 51 | 58 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 19 | 18 | 75
  >=65 years | 32 | 37 | 32 | 40 | 141
Age Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (7.2) | 68.6 (7.0) | 68.5 (7.2) | 69.1 (7.3) | 68.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 34 | 34 | 124
  Male | 22 | 29 | 17 | 24 | 92
Region of Enrollment [Number; unit: participants]
  United States | 51 | 56 | 51 | 58 | 216

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction Post-Vaccination 1.
Description: Solicited injection site reactions: pain, erythema, and swelling. Solicited systemic reactions: Fever (temperature), Headache, Malaise, Myalgia, chills, Arthralgia, Urticaria, Anorexia, Diarrhea, and Vomiting.
Time Frame: 0-7 days post-vaccination 1
Population: Safety analysis post-vaccination 1 was on all enrolled and vaccinated participants, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 51 | 56 | 51 | 58
Participants
  Any Solicited Injection Site Reaction | 26 | 20 | 28 | 23
  Grade 3 Solicited Injection Site Reaction | 4 | 0 | 1 | 3
  Any Pain | 12 | 16 | 24 | 18
  Grade 3 Pain (Incapacitating) | 1 | 0 | 0 | 1
  Any Erythema | 22 | 5 | 9 | 8
  Grade 3 Erythema (≥ 5 cm) | 3 | 0 | 1 | 0
  Any Swelling | 10 | 6 | 5 | 3
  Grade 3 Swelling (≥ 5 cm) | 0 | 0 | 1 | 2
  Any Solicited Systemic Reaction | 20 | 23 | 19 | 23
  Grade 3 Solicited Systemic Reaction | 3 | 1 | 3 | 3
  Any Anorexia | 3 | 4 | 1 | 2
  Grade 3 Anorexia (Prevents daily activities) | 2 | 0 | 1 | 0
  Any Arthralgia | 4 | 4 | 7 | 5
  Grade 3 Arthralgia (Prevents daily activities) | 1 | 0 | 2 | 2
  Any Chills | 4 | 4 | 1 | 1
  Grade 3 Chills (Prevents daily activities) | 1 | 0 | 0 | 1
  Any Diarrhea | 2 | 5 | 1 | 2
  Grade 3 Diarrhea (Prevents daily activities) | 0 | 0 | 0 | 0
  Any Fever | 3 | 2 | 0 | 3
  Grade 3 Fever (> 102.2 ºF) | 0 | 0 | 0 | 1
  Any Headache | 11 | 11 | 11 | 12
  Grade 3 Headache (Prevents daily activities) | 2 | 1 | 1 | 2
  Any Malaise | 6 | 6 | 5 | 9
  Grade 3 Malaise (Prevents daily activities) | 1 | 1 | 1 | 1
  Any Myalgia | 10 | 13 | 11 | 10
  Grade 3 Myalgia (Prevents daily activities) | 2 | 0 | 1 | 2
  Any Urticaria | 1 | 0 | 0 | 1
  Grade 3 Urticaria (Prevents daily activities) | 0 | 0 | 0 | 0
  Any Vomiting | 1 | 0 | 1 | 0
  Grade 3 Vomiting (Prevents daily activities) | 0 | 0 | 1 | 0

2. Other Pre Specified Outcome: Percentage of Participants With at Least a 4-fold Rise in Serum Bactericidal Antibody Titers Using Baby Rabbit Complement (SBA-BR) Post-Vaccination 1.
Time Frame: Day 28 Post-vaccination 1
Population: Serum bactericidal antibody titers using baby rabbit complement (SBA-BR) post-vaccination 1 were assessed in the per-protocol population. No data were collected for participants in Group 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 49 | 0 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A | 90 |  | 88 | 89
  Meningococcal Serogroup C | 86 |  | 68 | 75
  Meningococcal Serogroup Y | 84 |  | 56 | 54
  Meningococcal Serogroup W-135 | 92 |  | 51 | 73

3. Other Pre Specified Outcome: Percentage of Participants With at Least a 4-fold Rise in Serum Bactericidal Antibody Titers Using Baby Rabbit Complement (SBA-BR) Post-Vaccination 2
Time Frame: Day 28 Post-vaccination 2
Population: Serum bactericidal antibody titers using baby rabbit complement (SBA-BR) post-vaccination 2, were assessed in the per-protocol population. No data were collected for participants in Group 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 54 | 51 | 58
Percentage of Participants
  Meningococcal Serogroup A |  | 91 | 90 | 98
  Meningococcal Serogroup C |  | 72 | 85 | 83
  Meningococcal Serogroup Y |  | 66 | 76 | 73
  Meningococcal Serogroup W-135 |  | 72 | 73 | 81

4. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Serum Bactericidal Antibody Using Baby Rabbit Complement (SBA-BR) Pre- and Post-vaccination 1
Time Frame: Day 0 and Day 28 Post-vaccination 1
Population: Geometric mean titers of serum bactericidal antibody using baby rabbit complement (SBA-BR) pre- and post-vaccination 1 were assessed in the per-protocol population. No data were collected for participants in Group 2.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 49 | 0 | 41 | 48
Titers
  Meningococcal Serogroup A, Pre-dose 1 | 21.1 [11.0 to 40.5] |  | 18.6 [9.1 to 38.1] | 19.6 [10.0 to 38.3]
  Meningococcal Serogroup C, Pre-dose 1 | 9.9 [6.1 to 16.1] |  | 16.6 [8.5 to 32.2] | 7.6 [4.9 to 11.6]
  Meningococcal Serogroup Y, Pre-dose 1 | 27.4 [15.1 to 49.8] |  | 28.9 [14.9 to 56.0] | 14.9 [8.6 to 25.8]
  Meningococcal Serogroup W-135, Pre-dose 1 | 13.3 [8.0 to 22.0] |  | 10.3 [6.1 to 17.3] | 11.6 [7.1 to 19.2]
  Meningococcal Serogroup A, Post-dose 1 | 3870.7 [2611.0 to 5738.0] |  | 2048.0 [1082.2 to 3875.7] | 1874.6 [1199.7 to 2929.1]
  Meningococcal Serogroup C, Post-dose 1 | 927.5 [433.6 to 1983.8] |  | 529.6 [204.6 to 1370.9] | 367.3 [155.6 to 867.1]
  Meningococcal Serogroup Y, Post-dose 1 | 750.1 [434.8 to 1294.1] |  | 141.7 [63.5 to 316.3] | 143.7 [64.9 to 318.1]
  Meningococcal Serogroup W-135, Post-dose 1 | 782.7 [404.5 to 1514.4] |  | 78.4 [35.5 to 173.1] | 221.6 [117.4 to 418.1]

5. Post Hoc Outcome: Percentage of Participants With at Least a 4-fold Rise in Serum Bactericidal Antibody Titers Using Human Complement (SBA-HC) Post-vaccination 1
Time Frame: Day 28 Post-vaccination 1
Population: Serum bactericidal antibody using human complements (SBA-HC) titers post-vaccination 1 were determined in the per-protocol population. No data were collected for participants in Group 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 49 | 0 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A | 37 |  | 63 | 44
  Meningococcal Serogroup C | 31 |  | 44 | 35
  Meningococcal Serogroup Y | 49 |  | 20 | 29
  Meningococcal Serogroup W-135 | 47 |  | 20 | 33

6. Post Hoc Outcome: Percentage of Participants With at Least a 4-fold Rise in Serum Bactericidal Antibody Titers Using Human Complement (SBA-HC) Post-vaccination 2
Time Frame: 28 Days post-vaccination 2
Population: Serum bactericidal antibody using human complements (SBA-HC) titers post-vaccination 2 was determined in the per-protocol population. No data were collected for participants in Group 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 54 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A |  | 65 | 68 | 44
  Meningococcal Serogroup C |  | 48 | 44 | 48
  Meningococcal Serogroup Y |  | 48 | 29 | 40
  Meningococcal Serogroup W-135 |  | 44 | 27 | 46

7. Post Hoc Outcome: Geometric Mean Titers of Serum Bactericidal Antibody Using Human Complement (SBA-HC) Pre- and Post-vaccination 1
Time Frame: Day 0 and Day 28 Post-vaccination 1
Population: Geometric mean of serum bactericidal antibody titers using human complements (SBA-HC) pre- and post-vaccination 1 were determined in the per-protocol population. No data were collected for participants in Group 2.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 49 | 0 | 41 | 48
Titers
  Meningococcal Serogroup A, Pre-dose 1 | 4.6 [3.5 to 6.0] |  | 4.3 [3.3 to 5.6] | 4.1 [3.1 to 5.3]
  Meningococcal Serogroup C, Pre-dose 1 | 3.9 [2.9 to 5.4] |  | 3.1 [2.3 to 4.2] | 3.4 [2.6 to 4.5]
  Meningococcal Serogroup Y, Pre-dose 1 | 5.2 [3.4 to 7.9] |  | 3.4 [2.3 to 4.9] | 3.3 [2.4 to 4.4]
  Meningococcal Serogroup W-135, Pre-dose 1 | 2.8 [2.3 to 3.4] |  | 2.8 [2.3 to 3.4] | 3.1 [2.4 to 4.0]
  Meningococcal Serogroup A, Post-dose 1 | 14.3 [8.8 to 23.1] |  | 40.5 [20.3 to 80.8] | 22.6 [13.0 to 39.4]
  Meningococcal Serogroup C, Post-dose 1 | 15.1 [8.2 to 27.8] |  | 18.9 [9.2 to 38.9] | 14.9 [7.7 to 28.8]
  Meningococcal Serogroup Y, Post-dose 1 | 23.8 [12.8 to 44.2] |  | 6.8 [4.0 to 11.4] | 10.4 [5.9 to 18.3]
  Meningococcal Serogroup W-135, Post-dose 1 | 13.5 [8.6 to 21.1] |  | 7.1 [4.3 to 11.8] | 12.5 [6.7 to 23.2]

8. Primary Outcome: Number of Participants With At Least One Solicited Injection Site Reaction Post-Vaccination 2
Description: Solicited injection site reactions: Pain, Erythema, and Swelling.
Time Frame: 0-7 Days Post-vaccination 2
Population: Safety analysis post-vaccination 2 was on all enrolled and vaccinated participants, intent-to-treat population. No data were collected for participants in Group 1.
Measure: Number; unit: Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 56 | 51 | 58
Participants
  Any Solicited Injection site reaction |  | 17 | 25 | 24
  Grade 3 Solicited Injection site reaction |  | 0 | 0 | 1
  Any Pain |  | 14 | 24 | 22
  Grade 3 Pain (Incapacitating) |  | 0 | 0 | 0
  Any Erythema |  | 7 | 5 | 6
  Grade 3 Erythema (≥ 5 cm) |  | 0 | 0 | 1
  Any Swelling |  | 5 | 5 | 3
  Grade 3 Swelling (≥ 5 cm) |  | 0 | 0 | 1

9. Primary Outcome: Number of Participants With At Least One Solicited Systemic Reaction Post-Vaccination 2
Description: Solicited systemic reactions: Fever (temperature), Headache, Malaise, Myalgia, chills, Arthralgia, Urticaria, Anorexia, Diarrhea, and Vomiting.
Time Frame: Day 0 to 7 Post-vaccination 2
Population: Safety analysis post-vaccination 2 was on all enrolled and vaccinated participants, intent-to-treat population. No data were collected for participants in Group 1 and Group 2.
Measure: Number; unit: Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 0 | 51 | 58
Participants
  Any Solicited Systemic Reaction |  |  | 19 | 13
  Grade 3 Solicited Systemic Reaction |  |  | 3 | 1
  Any Anorexia |  |  | 1 | 2
  Grade 3 Anorexia (Prevents daily activities) |  |  | 0 | 0
  Any Arthralgia |  |  | 5 | 2
  Grade 3 Arthralgia (Prevents daily activities) |  |  | 1 | 2
  Any Chills |  |  | 4 | 1
  Grade 3 Chills (Prevents daily activities) |  |  | 0 | 1
  Any Diarrhea |  |  | 2 | 3
  Grade 3 Diarrhea (Prevents daily activities) |  |  | 0 | 0
  Any Fever |  |  | 0 | 3
  Grade 3 Fever (> 102.2 ºF) |  |  | 0 | 1
  Any Headache |  |  | 9 | 7
  Grade 3 Headache (Prevents daily activities) |  |  | 1 | 2
  Any Malaise |  |  | 10 | 3
  Grade 3 Malaise (Prevents daily activities) |  |  | 0 | 1
  Any Myalgia |  |  | 12 | 7
  Grade 3 Myalgia (Prevents daily activities) |  |  | 0 | 2
  Any Urticaria |  |  | 1 | 0
  Grade 3 Urticaria (Prevents daily activities) |  |  | 0 | 0
  Any Vomiting |  |  | 0 | 0
  Grade 3 Vomiting (Prevents daily activities) |  |  | 0 | 0

10. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Serum Bactericidal Antibody Using Baby Rabbit Complement (SBA-BR) Pre-vaccination 1 and Post-vaccination 2
Time Frame: Day 0 and 28 days Post-vaccination 2
Population: Geometric mean titers of serum bactericidal antibody using baby rabbit complement pre-vaccination 1 and post-vaccination 2 was determined in per-protocol population. No data were collected for participants in Group 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 54 | 41 | 48
Titers
  Meningococcal Serogroup A, Pre-dose 1 |  | 16.8 [8.7 to 32.5] | 18.6 [9.1 to 38.1] | 19.6 [10.0 to 38.3]
  Meningococcal Serogroup C, Pre-dose 1 |  | 11.0 [6.5 to 18.6] | 16.6 [8.5 to 32.2] | 7.6 [4.9 to 11.6]
  Meningococcal Serogroup Y, Pre-dose 1 |  | 22.6 [14.2 to 36.1] | 28.9 [14.9 to 56.0] | 14.9 [8.6 to 25.8]
  Meningococcal Serogroup W-135, Pre-dose 1 |  | 12.9 [7.4 to 22.2] | 10.3 [6.1 to 17.3] | 11.6 [7.1 to 19.2]
  Meningococcal Serogroup A, Post-dose 2 |  | 3168.6 [2056.7 to 4881.7] | 2871.9 [1823.9 to 4522.1] | 2543.3 [1791.8 to 3610.0]
  Meningococcal Serogroup C, Post-dose 2 |  | 568.5 [240.0 to 1346.2] | 1041.5 [492.4 to 2202.9] | 574.7 [251.7 to 1312.1]
  Meningococcal Serogroup Y, Post-dose 2 |  | 311.5 [173.4 to 559.5] | 264.8 [135.7 to 516.9] | 259.7 [128.0 to 527.0]
  Meningococcal Serogroup W-135, Post-dose 2 |  | 276.9 [135.1 to 567.4] | 212.6 [96.3 to 469.2] | 566.5 [299.3 to 1071.9]

11. Other Pre Specified Outcome: Percentage of Participants Achieving Serum Bactericidal Antibody Using Baby Rabbit Complement (SBA-BR) Titers of at Least 1:8 (≥1:8) Pre- and Post-vaccination 1
Time Frame: Day 28 Post-vaccination 1
Population: Serum bactericidal antibody titers using baby rabbit complement (SBA-BR) pre- and post-vaccination 1 were assessed in the per-protocol population. No data were collected for participants in Group 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 49 | 0 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A ≥ 1:8 Pre-Dose 1 | 38 |  | 34 | 35
  Meningococcal Serogroup C ≥ 1:8 Pre-Dose 1 | 25 |  | 34 | 19
  Meningococcal Serogroup Y ≥1:8 Pre-Dose 1 | 55 |  | 54 | 38
  Meningococcal Serogroup W-135 ≥ 1:8 Pre-Dose 1 | 35 |  | 29 | 33
  Meningococcal Serogroup A ≥ 1:8 Post-Dose 1 | 100 |  | 95 | 98
  Meningococcal Serogroup C ≥ 1:8 Post-Dose 1 | 88 |  | 78 | 79
  Meningococcal Serogroup Y ≥ 1:8 Post-Dose 1 | 96 |  | 78 | 71
  Meningococcal Serogroup W-135 ≥ 1:8 Post-Dose 1 | 94 |  | 68 | 90

12. Other Pre Specified Outcome: Percentage of Participants Achieving Serum Bactericidal Antibody Using Baby Rabbit Complement (SBA-BR) Titers of at Least 1:8 (≥1:8), Pre-vaccination 1 and Post-vaccination 2
Time Frame: Day 0 and Day 28 Post-vaccination 2
Population: Serum bactericidal antibody using baby rabbit complement titer pre-vaccination 1 and post-vaccination 2 were determined in the per-protocol population. No data were collected for participants in Group 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 54 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A, ≥ 1:8 Pre-dose 1 |  | 28 | 34 | 35
  Meningococcal Serogroup C, ≥ 1:8 Pre-dose 1 |  | 24 | 34 | 19
  Meningococcal Serogroup Y, ≥ 1:8 Pre-dose 1 |  | 54 | 54 | 38
  Meningococcal Serogroup W-135, ≥ 1:8 Pre-dose 1 |  | 30 | 29 | 33
  Meningococcal Serogroup A, ≥ 1:8 Post-dose 2 |  | 98 | 100 | 100
  Meningococcal Serogroup C, ≥ 1:8 Post-dose 2 |  | 79 | 90 | 83
  Meningococcal Serogroup Y, ≥ 1:8 Post-dose 2 |  | 93 | 90 | 85
  Meningococcal Serogroup W-135, ≥ 1:8 Post-dose 2 |  | 83 | 81 | 94

13. Post Hoc Outcome: Geometric Mean Titers of Serum Bactericidal Antibody Using Human Complement (SBA-HC) Pre-vaccination 1 and Post-vaccination 2
Time Frame: Day 0 and Day 28 Post-vaccination 2
Population: Geometric mean of serum bactericidal antibody titers using human complement (SBA-HC) pre-vaccination 1 and post-vaccination 2 were determined in the per-protocol population. No data were collected for participants in Group 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 56 | 51 | 58
Titers
  Meningococcal Serogroup A, Pre-dose 1 |  | 4.9 [3.5 to 6.9] | 4.3 [3.3 to 5.6] | 4.1 [3.1 to 5.3]
  Meningococcal Serogroup C, Pre-dose 1 |  | 3.9 [2.9 to 5.3] | 3.1 [2.3 to 4.2] | 3.4 [2.6 to 4.5]
  Meningococcal Serogroup Y Pre-dose 1 |  | 5.4 [3.8 to 7.7] | 3.4 [2.3 to 4.2] | 3.3 [2.4 to 4.4]
  Meningococcal Serogroup W-135, Pre-dose 1 |  | 4.3 [3.1 to 5.8] | 2.8 [2.3 to 3.4] | 3.1 [2.4 to 4.0]
  Meningococcal Serogroup A, Post-dose 2 |  | 47.6 [26.9 to 84.2] | 48.0 [27.4 to 84.2] | 21.1 [12.6 to 35.0]
  Meningococcal Serogroup C, Post-dose 2 |  | 25.7 [13.8 to 47.9] | 17.7 [8.9 to 35.3] | 18.8 [9.9 to 35.6]
  Meningococcal Serogroup Y, Post-dose 2 |  | 28.1 [16.0 to 49.6] | 10.1 [5.7 to 18.0] | 12.7 [7.3 to 22.1]
  Meningococcal Serogroup W-135, Post-dose 2 |  | 26.1 [14.0 to 48.5] | 9.3 [5.5 to 15.7] | 18.2 [10.3 to 32.3]

14. Post Hoc Outcome: Percentage of Participants Achieving Serum Bactericidal Antibody Using Human Complement (SBA-HC) Titers of at Least 1:8 (≥1:8) Pre- and Post-vaccination 1.
Time Frame: Day 28 Post-vaccination 1
Population: Serum bactericidal antibody using human complement (SBA-HC) titers pre- and post-vaccination 1 were determined in the per-protocol population. No data were collected for participants in Group 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 49 | 0 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A, Pre-dose 1 | 39 |  | 32 | 27
  Meningococcal Serogroup C, Pre-dose 1 | 22 |  | 15 | 19
  Meningococcal Serogroup Y, Pre-dose 1 | 31 |  | 17 | 17
  Meningococcal Serogroup W-135, Pre-dose 1 | 16 |  | 12 | 19
  Meningococcal Serogroup A, Post-dose 1 | 63 |  | 76 | 73
  Meningococcal Serogroup C, Post-dose 1 | 57 |  | 56 | 52
  Meningococcal Serogroup Y, Post-dose 1 | 63 |  | 37 | 44
  Meningococcal Serogroup W-135, Post-dose 1 | 63 |  | 46 | 50

15. Post Hoc Outcome: Percentage of Participants Achieving Serum Bactericidal Antibody Using Human Complement (SBA-HC) Titers of at Least 1:8 (≥1:8) Pre-vaccination 1 and Post-vaccination 2
Time Frame: Day 0 and 28 days post-vaccination
Population: Serum bactericidal antibody using human complement (SBA-HC) pre-vaccination 1 and post-vaccination 2 were determined in the per-protocol population. No data were collected for participants in Group 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menomune® Day 0 | Group 2: Menactra® Day 0 x 2 | Group 3: Menactra® Day 0 and 14 | Group 4: Menactra® Day 0 and 28
Number analyzed (Participants) | 0 | 54 | 41 | 48
Percentage of Participants
  Meningococcal Serogroup A, Pre-dose 1 |  | 33 | 32 | 27
  Meningococcal Serogroup C, Pre-dose 1 |  | 22 | 15 | 19
  Meningococcal Serogroup Y, Pre-dose 1 |  | 37 | 17 | 17
  Meningococcal Serogroup W-135, Pre-dose 1 |  | 26 | 12 | 19
  Meningococcal Serogroup A, Post-dose 2 |  | 82 | 81 | 75
  Meningococcal Serogroup C, Post-dose 2 |  | 65 | 56 | 65
  Meningococcal Serogroup Y, Post-dose 2 |  | 72 | 54 | 54
  Meningococcal Serogroup W-135, Post-dose 2 |  | 63 | 56 | 63

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from day of enrollment to 6 Months after the last vaccination.
Arm/Group | Menomune® Day 0 | Menactra® Day 0 x 2 | Menactra® Day 0 and Day 14 | Menactra® Day 0 and Day 28
Serious Adverse Events (participants affected / at risk) | 4/51 | 3/56 | 1/51 | 0/58
Other Adverse Events (participants affected / at risk) | 3/51 | 5/56 | 8/51 | 12/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menomune® Day 0 (N=51) | Menactra® Day 0 x 2 (N=56) | Menactra® Day 0 and Day 14 (N=51) | Menactra® Day 0 and Day 28 (N=58)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus non-insulin-dependent (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menomune® Day 0 (N=51) | Menactra® Day 0 x 2 (N=56) | Menactra® Day 0 and Day 14 (N=51) | Menactra® Day 0 and Day 28 (N=58)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 2 (2) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 2 (2) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications